CLINICAL TRIAL: NCT06437717
Title: Role of Nanoemulsified Sesame Oil in Post-operative Care After Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha A.Elkholy, Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.20.5.1134
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-05

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- only normal saline as nasal irrigation (Active Comparator)
  Interventions: Other: application of different topical nasal solutions
- normal saline as nasal irrigation followed by sesame oil nasal drops (Active Comparator)
  Interventions: Other: application of different topical nasal solutions
- only Ringer's lactate solution as nasal irrigation (Active Comparator)
  Interventions: Other: application of different topical nasal solutions
- Ringer's lactate solution as nasal irrigation followed by sesame oil nasal drops (Active Comparator)
  Interventions: Other: application of different topical nasal solutions

INTERVENTIONS:
Other: application of different topical nasal solutions — each group receives a type of nasal solution to detect if there is a difference in the outcomes in chronic rhinosinusitis patients

SUMMARY:
The goal of our thesis is to design, develop and characterize a novel thermodynamically stable NE by spontaneous method intended for topical use. Subsequently, appraisal of nanoemulsified sesame oil formulation has been performed on the post-operative symptoms in CRS patients who have undergone ESS (endoscopic sinus surgery) combined with different types of nasal irrigation which may affect formulation efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age between 18 and 60 years old.
2. chronic rhinosinusitis patients who have undergone endoscopic sinus surgery.

Exclusion Criteria:

1. Patients with history of allergy for sesame seed derivatives.
2. Patients with chronic diseases which affecting the process of healing (uncontrolled DM, renal failure and hepatic failure).
3. Patients with nasal granulomas.
4. Patients with invasive fungal rhinosinusitis.
5. Smokers.
6. Patients with history of radio and/or chemotherapy exposure.
7. Patients with systemic diseases affecting integrity of nasal mucosa (e.g. CF, scleroderma, Sjogren syndrome …).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Sinonasal Outcome Test 22 (SNOT-22) | weekly for three months
Lund-Kennedy endoscopic grading system | once monthly for three months

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: No